CLINICAL TRIAL: NCT04522830
Title: A Double-blind, Placebo-controlled, Phase 2 Trial of Sublingual Low-Dose Thimerosal in Adults With Symptomatic SARS-CoV-2 Infection
Brief Title: A Study in Adults to Test the Effects of Low Dose Thimerosal on Symptoms of COVID-19
Acronym: BTL-TML-COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beech Tree Labs, Inc. (Industry)
Collaborators: Norwich Clinical Research Associates Ltd. (Other); Curavit Clinical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-04-0311
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: SARS-CoV-2 Infection
Keywords: Treatment for COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BTL-TML-COVID (Experimental): BTL-TML-COVID
  Interventions: Drug: BTL-TML-COVID
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BTL-TML-COVID — Sublingual dosing of BTL-TML-COVID on days 1 and 2 - Day 1 - 1 drop every 15 minutes for the first hour of initiation of treatment then every hour for the balance of the day until bedtime.
  Day 2 - 1 drop every 2-3 hours for a total of 6 times during the day. The parallel group assignment will only be maintained until the completion of a minimum of 48 hours of blinded study drug dosing, at which point all subjects will receive the active treatment.
  Day 3 - 1 drop every 15 mins for the first hour of the day, then every hour for the balance of the day until bedtime.
  Days 4 through 10 - 1 drop every 3-4 hours for a total of four times during the day.
  Arms: BTL-TML-COVID
Drug: Placebo — Sublingual dosing of matching placebo on days 1 and 2 - Day 1 - 1 drop every 15 minutes for the first hour of initiation of treatment then every hour for the balance of the day until bedtime.
  Day 2 - 1 drop every 2-3 hours for a total of 6 times during the day. The parallel group assignment will only be maintained until the completion of a minimum of 48 hours of blinded study drug dosing, at which point all subjects will receive the active treatment.
  Day 3 - 1 drop every 15 mins for the first hour of the day, then every hour for the balance of the day until bedtime.
  Days 4 through 10 - 1 drop every 3-4 hours for a total of four times during the day.
  Arms: Placebo

SUMMARY:
Clinical trial to compare sublingual low does thimerosal in adults that have symptoms of SARS-CoV-2 Infection against placebo to show a difference in physical characteristics and viral levels.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older
* Provide written informed consent
* Have a SARS-COV-19 diagnostic test with positive results

Exclusion Criteria:

* Having an oxygen saturation level below 92% at baseline or currently on Oxygen therapy
* Subjects currently hospitalized
* Subjects who have received a COVID vaccination
* Subjects with a diagnosis of immunodeficiency

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Mean duration and severity of disease | Two days
  Change from baseline in the physical component summary of the short form-36 Quality of Life Instrument

SECONDARY OUTCOMES:
Incidence/Safety of Adverse Events | Baseline through 10 days
  AEs will be assessed by the investigator as to severity, duration and relationship to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Duane Harris, MD, Principal Investigator — Intermountain Clinical Research; Lee Truax-Bellows, Study Director — Norwich Clinical Research Associates (NCRA)
Locations (1):
- Intermountain Clinical Reserach, Draper, Utah, United States

IPD SHARING:
Plan to Share IPD: No